CLINICAL TRIAL: NCT04544319
Title: Clinical Trial to Compare the Pharmacokinetics, Safety and Tolerability of the FDC of Gemigliptin/Dapagliflozin 50/10 mg to Each Component of Gemigliptin 50 mg and Dapagliflozin 10 mg
Brief Title: Clinical Trial to Compare the PK of the Fixed-dose Combinations and Each Component of Gemigliptin/Dapagliflozin 50/10 mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-GLCL002
Record Dates: First submitted 2020-07-29; First posted 2020-09-10 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: T2DM
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Firstly, administrating each component Gemigliptin 50mg and dapagliflozin 10mg and after resting period administrating Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg
  Interventions: Drug: Zemiglo 50mg and Forxiga 10mg; Drug: Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg
- Arm II (Experimental): Firstly, administrating Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg and after resting period administrating each component Gemigliptin 50mg and dapagliflozin 10mg
  Interventions: Drug: Zemiglo 50mg and Forxiga 10mg; Drug: Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg

INTERVENTIONS:
Drug: Zemiglo 50mg and Forxiga 10mg — Each component of Gemigliptin 50mg QD and Dapagliflozin 10mg QD
  Other Names: zemiglo and Forxiga
Drug: Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg — Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg QD
  Other Names: zemiglo and Forxiga

SUMMARY:
To identify bioequivalence between Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg to Each Component of Gemigliptin 50 mg and Dapagliflozin 10 mg

DETAILED DESCRIPTION:
To identify bioequivalence between Fixed-dose Combinations of Gemigliptin/Dapagliflozin 50/10 mg and each Component of Gemigliptin 50 mg and Dapagliflozin 10 mg Also we identify safety and tolerance of FDC and each component

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults who are 19 years ~ 50 years when they are screened
2. weight: 55.0 kg ~ 90.0 kg and BMI: 18.0 kg/m2 ~ 30.0 kg/m2
3. Volunteers who understand the procedures of clinical trial and signed informed consent form
4. Volunteers who are eligible decided by vital signs, physical examination, lab test and 12-lead ECG
5. Women of chlidbearing potential have negative results in pregnancy test

Exclusion Criteria:

1. Healtjy volunteers who don't have clinically significant disease such as liver disease, severe renal disease, acute pancreatitis... etc
2. Drug Allergy in aspirin, NSAID, Anti-bacterial drugs
3. GI tract diseases which affect PK results and safety such as ulceritis, GERD, chron disease...
4. Chronic urine track infection
5. Allergy history in sunset yellow 5 pigment and Fast green FCF (pigment)
6. galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
7. These resluts are appeared when screening

   * ALT, AST >= 1.5 Upper limit of normal range
   * HbsAg, anti-HCV, HIV Ag&Ab positive
   * MDRD equation: eGFR< 60 mL/min/1.73m2
   * QTcB> 450 ms
   * Fasting serum glucose < 70mg/dL or >110mg/dL
   * HbA1c>6.5%
8. SBP<90mmHg or >150mmHg, DBP <60mmHg or >100mmHg

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Gemigliptin and dapagliflozin AUClast and Cmax | Pre-dose (Day1 0 hour)
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 0.25hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 0.5hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 0.75hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 1hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 1.5hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 2hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 3hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 4hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 6hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 8hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 10hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 12hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 24hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 36hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 48hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin AUClast and Cmax | Day 1 72hour
  each phase 17 times blood sampling, total 34 times blood sampling

SECONDARY OUTCOMES:
Gemigliptin and dapagliflozin AUCinf | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin Tmax | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin t1/2 | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin CL/F | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin and dapagliflozin V/F | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin metabolite(LC15-0636) AUClast | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin metabolite(LC15-0636) Cmax | Pre-dose (Day1 0 h), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin metabolite(LC15-0636) AUCinf | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin metabolite(LC15-0636) t1/2 | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling
Gemigliptin metabolite(LC15-0636) metabolic ratio | Pre-dose (Day1 0 hour), Day 1 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  each phase 17 times blood sampling, total 34 times blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: seunghwan Lee, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No